CLINICAL TRIAL: NCT07110324
Title: Characteristics of Persistent Pain Composition Following Total Hip or Knee Arthroplasty: a Descriptive Study
Acronym: PAIN-COMPO
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Milan Mohammad, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: 20042025PAINCOMPO
Record Dates: First submitted 2025-06-26; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Pain (Visceral, Somatic, or Neuropathic); Hip Arthroplasty Replacement; Knee Arthroplasty, Total; Survey and Questionnaire
Keywords: Pain; hip arthroplasty; knee arthroplasty
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persistant pain (NRS above 3): Explore the pain composition in terms of neuropathic, nociceptive and nociplastic pain in patients with persistent pain after total knee arthroplasty (TKA), total hip arthroplasty (THA), or unicompartmental knee arthroplasty (UKA).

SUMMARY:
Despite high success rates of hip and knee arthroplasty, up to 20% of patients report moderate-to-severe pain (NRS > 3) persisting beyond the expected healing period. This investigator-initiated, descriptive cohort study will re-invite approximately 100 consenting patients with persistent postoperative pain-identified from a pool of ~7 000 respondents-to complete standardized assessments of neuropathic (DN4), nociplastic (IASP criteria + Fibromyalgia Survey Questionnaire) and nociceptive (KOOS/HOOS pain domains) pain. Primary outcomes are the prevalence of potential nociplastic pain and the proportion experiencing significant pain in two or more mechanistic categories. Secondary analyses will compare baseline vs. re-evaluated DN4 scores, FSQ and KOOS/HOOS distributions, and examine differences between patients with and without possible neuropathic pain. Findings will inform targeted pre- and postoperative pain management strategies.

DETAILED DESCRIPTION:
Introduction Background: Knee and hip arthroplasties are primarily performed due to degenerative changes that typically result in pain, functional impairment, and a subsequent decline in quality of life [1]. Arthroplasty represents the definitive intervention, involving the removal of the degenerated, pain-inducing joint components and their replacement with artificial prostheses. These procedures are considered standard in orthopedic surgery, boasting high success rates and high levels of patient satisfaction [2,3,4]. Nevertheless, the surgeries are not without risks, including perioperative complications such as infection, thrombosis, and prosthetic dislocation. Additionally, the economic burden on healthcare systems is considerable, encompassing not only the costs of the surgery itself but also postoperative care and rehabilitation. Hence, it is essential that the procedure yields the desired pain-relieving and functional outcomes to justify its use. Osteoarthritis is the primary indication for arthroplasty, representing a leading cause of disability worldwide. In advanced stages of osteoarthritis, the pain profile can become multifaceted, often involving a combination of nociceptive, neuropathic, and nociplastic pain mechanisms. Nociceptive pain, stemming from joint tissue damage and inflammation, is the most prevalent form and is usually effectively managed by arthroplasty. However, the complexity of pain perception in osteoarthritis extends beyond the joint, potentially involving altered pain processing pathways within the central and peripheral nervous systems. Up to 20% of patients report significant persistent pain following arthroplasty despite uncomplicated surgery and no apparent source of pain. This could be explained by the presence of non-nociceptive pain. Neuropathic pain stem from nerve damage, while nociplastic pain is associated with altered central pain processing, leading to pain persisting even after the natural healing process [5]. Identifying the type of pain in patients with persistent post-surgical pain could have important implications for pre-surgical as well as post-surgical management.

Objective: The aim of this study is to explore the pain composition in terms of neuropathic, nociceptive and nociplastic pain in patients with persistent pain after total knee arthroplasty (TKA), total hip arthroplasty (THA), or unicompartmental knee arthroplasty (UKA).

Hypotheses: The investigators hypothesize that postoperative pain with multiple pain types is prevalent and that neuropathic and nociplastic pain is co-existent or conflated in a considerable proportion of patients. Thus, there is an increased prevalence of potential nociplastic pain among patients with a Neuropathic Pain score (DN4) reflecting 'possible neuropathic pain'.

Perspective: Correct identification of pain types has important implications for pain management pre-operatively, peri-operatively, and post-operatively. Moreover, a high proportion of patients with potential nociplastic pain could increase the focus on the link between preoperative patient characteristics and post-operative potential nociplastic pain. This would help targeting those individuals benefiting most from operation compared to non-surgical management. Although results from this post-operative population do not necessarily reflect the prevailing pre-operative pain composition, the results from the study can potentially form the basis for hypothesis testing in a pre-operative cohort.

Methods This protocol was registered before initiation of data collection.

Study design Descriptive Cohort Study: Approximately 7,000 patients have been administered questionnaires to indicate persistent postoperative pain including the DN4 questionnaire to indicate potential neuropathic pain [6]. All patients with evidence of persistent pain following operation and have consented to be contacted, will receive invitation to participate in the study to complete new patient-reported outcome measures (PROMs). For comparison in pain composition between patients with and without possible neuropathic pain, the investigators expect to include 100 patients with possible neuropathic pain, as around 6% of the 7,000 (with 25% consenting to be contacted) scored high enough to consider possible neuropathic pain.

Variables The DN4 will be administered again to assess any development. Nociplastic pain will be evaluated based on the International Association for the Study of Pain (IASP) criteria and using the Fibromyalgia Survey Questionnaire (FSQ), and nociceptive pain will be measured through Knee injury and Osteoarthritis Outcome Pain Domain Score (KOOS) / Hip Disability and Osteoarthritis Outcome Score (HOOS). Patients will also be asked about their satisfaction with the outcome and their thoughts on potential re-operation.

Outcomes

* Primary outcomes: Prevalence of potential nociplastic pain (defined by IASP criteria) and proportion of patients with significant painscores in two or more pain categories.
* Secondary outcomes:

  1. Difference between baseline and re-evaluated DN4i (DN4 interview) score.
  2. Prevalence of potential nociplastic pain, as assessed with the FSQ score.
  3. Distribution of KOOS/HOOS score.
  4. Difference in pain distribution in terms of IASP, FSQ, KOOS / HOOS in patients with possible neuropathic pain (DN4 score above 3) and patients without any kind of neuropathic pain (DN4 score equal to zero). (Substudy)
* Exploratory: The investigators explore rates of satisfaction and consideration of re-operation.

Inclusion and exclusion criteria:

Inclusion criteria: All patients with persistent moderate-severe pain (NRS>3) after THA, TKA and UKA and acceptance to be contacted.

Exclusion criteria: Re-operation or luxation, do not want to be contacted, post-operative complications such as prosthesis infection, thromboembolism or fracture of the prosthesis.

Questionnaires

The questionnaire is a combination of following questionnaires (Appendix A):

* DN4: To assess the presence of neuropathic pain, the DN4 questionnaire will be administered. This tool evaluates symptoms and characteristics of pain that may indicate neuropathic origins [7].
* Nociplastic Pain Assessment: Based on the new IASP diagnostic criteria for complex regional pain syndrome (CRPS) (aka "the Budapest Criteria), patients will be assessed for nociplastic pain, which involves pain arising from altered pain processing [8].
* KOOS/HOOS: The pain domain of the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Hip Disability and Osteoarthritis Outcome Score (HOOS) will be used to measure nociceptive pain and overall functional outcomes in the knee and hip joints, respectively ([9,10]. Scores ranges from 100 (equal to no pain) 0 (extreme pain). A score equal to or below 60 is considered significant.
* Fibromyalgia Survey Questionnaire (FSQ): This questionnaire will also be used to identify symptoms consistent with nociplastic pain, which can mimic or coexist with postoperative pain [11]. A score equal to or greater than 13 points is consistent with a diagnosis of fibromyalgia, the most common nociplastic pain condition.
* Satisfaction and re-operation: Patients will be queried about their satisfaction with the surgical outcome and their thoughts on the possibility of undergoing additional surgical interventions.

Statistical considerations

Descriptive cohort study. As such, no formal power calculation is conducted and the sample size depends on response rate form an pre-defined cohort. All statistical analyses will be conducted by using R statistical software version 4.1.1 (R Foundation for Statistical Computing, Vienna, Austria). within RStudio (version 1.4.1717). A two-tailed P < 0.05 will be considered statistically significant. Data will be reported as mean (standard deviation (SD)) and mean difference (95% confidence interval (95% CI): lower limit (LL), upper limit (UL)).

References:

1. Wiklund I, Romanus B. A comparison of quality of life before and after arthroplasty in patients who had arthrosis of the hip joint. J Bone Joint Surg Am. 1991 Jun;73(5):765-9. PMID: 2045402.
2. Papakostidou I, Dailiana ZH, Papapolychroniou T, Liaropoulos L, Zintzaras E, Karachalios TS, Malizos KN. Factors affecting the quality of life after total knee arthroplasties: a prospective study. BMC Musculoskelet Disord. 2012 Jun 29;13:116. doi: 10.1186/1471-2474-13-116. PMID: 22748117; PMCID: PMC3476961.
3. Snell DL, Dunn JA, Hooper G. Associations between pain, function and quality of life after total hip arthroplasty. Int J Orthop Trauma Nurs. 2024 Aug;54:101121. doi: 10.1016/j.ijotn.2024.101121. Epub 2024 Jul 14. PMID: 39029151.
4. Shapira J, Chen SL, Rosinsky PJ, Maldonado DR, Lall AC, Domb BG. Outcomes of outpatient total hip arthroplasty: a systematic review. HIP International. 2021;31(1):4-11. doi:10.1177/1120700020911639
5. Soni A, Wanigasekera V, Mezue M, Cooper C, Javaid MK, Price AJ, Tracey I. Central Sensitization in Knee Osteoarthritis: Relating Presurgical Brainstem Neuroimaging and PainDETECT-Based Patient Stratification to Arthroplasty Outcome. Arthritis Rheumatol. 2019 Apr;71(4):550-560. doi: 10.1002/art.40749. Epub 2019 Mar 6. PMID: 30295432; PMCID: PMC6430421.
6. Bennett, M. I., Attal, N., Backonja, M. M., Baron, R., Bouhassira, D., Freynhagen, R., Scholz, J., Tölle, T. R., Wittchen, H. U., & Jensen, T. S. (2007). Using screening tools to identify neuropathic pain. Pain, 127(3), 199-203.
7. Spallone, V., Morganti, R., D'Amato, C., Greco, C., Cacciotti, L., & Marfia, G. A. (2012). Validation of DN4 as a screening tool for neuropathic pain in painful diabetic polyneuropathy. Diabetic medicine : a journal of the British Diabetic Association, 29(5), 578-585.
8. Goebel A, Birklein F, Brunner F, Clark JD, Gierthmühlen J, Harden N, Huygen F, Knudsen L, McCabe C, Lewis J, Maihöfner C, Magerl W, Moseley GL, Terkelsen A, Thomassen I, Bruehl S. The Valencia consensus-based adaptation of the IASP complex regional pain syndrome diagnostic criteria. Pain. 2021 Sep 1;162(9):2346-2348.
9. Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64.
10. Nilsdotter, A. K., Lohmander, L. S., Klässbo, M., & Roos, E. M. (2003). Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC musculoskeletal disorders, 4, 10.
11. Häuser, W., Jung, E., Erbslöh-Möller, B., Gesmann, M., Kühn-Becker, H., Petermann, F., Langhorst, J., Weiss, T., Winkelmann, A., & Wolfe, F. (2012). Validation of the Fibromyalgia Survey Questionnaire within a cross-sectional survey. PloS one, 7(5), e37504. https://doi.org/10.1371/journal.pone.0037504

ELIGIBILITY:
Inclusion Criteria:

* All patients with persistent moderate-severe pain (NRS>3) after THA, TKA and UKA
* Acceptance to be contacted.

Exclusion Criteria:

* Re-operation
* Luxation
* Do not want to be contacted
* Post-operative complications such as prosthesis infection, thromboembolism or fracture of the prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Descriptive Cohort Study: Approximately 7,000 patients have been administered questionnaires to indicate persistent postoperative pain including the DN4 questionnaire to indicate potential neuropathic pain [6]. All patients with evidence of persistent pain following operation and have consented to be contacted, will receive invitation to participate in the study to complete new patient-reported outcome measures (PROMs). For comparison in pain composition between patients with and without possible neuropathic pain, we expect to include 100 patients with possible neuropathic pain, as around 6% of the 7,000 (with 25% consenting to be contacted) scored high enough to consider possible neuropathic pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Potential nociplastic pain | 1 year
  Prevalence of potential nociplastic pain (defined by International Association for the Study of Pain criteria)

SECONDARY OUTCOMES:
Difference between baseline and re-evaluated neuropathic pain score. | 1 year
  Difference between baseline and re-evaluated neuropathic pain score.
Prevalence of potential nociplastic pain, as assessed with the Fibromyalgia Survey Questionnaire score. | 1 year
  Prevalence of potential nociplastic pain, as assessed with the Fibromyalgia Survey Questionnaire score.
Distribution of Knee injury and Osteoarthritis Outcome Score (KOOS) | 1 year
  Distribution of Knee injury and Osteoarthritis Outcome Score (KOOS)
Distribution of Hip injury and Osteoarthritis Outcome Score (HOOS) | 1 year
  Distribution of Hip injury and Osteoarthritis Outcome Score (HOOS)

OTHER OUTCOMES:
Difference in pain distribution in terms of International Association for the Study of Pain score in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero). | 1 year
  Difference in pain distribution in terms of International Association for the Study of Pain score in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero).
Rates of satisfaction | 1 year
  Rates of satisfaction
Rates of consideration of re-operation. | 1 year
  Rates of consideration of re-operation.
Difference in pain distribution in terms of Fibromyalgia Survey Questionnaire score in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero). | 1 year
  Difference in pain distribution in terms of Fibromyalgia Survey Questionnaire score in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero).
Difference in pain distribution in terms of Knee injury and Osteoarthritis Outcome Score (KOOS) in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero). | 1 year
  Difference in pain distribution in terms of Knee injury and Osteoarthritis Outcome Score (KOOS) in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero).
Difference in pain distribution in terms of Hip injury and Osteoarthritis Outcome Score (HOOS) in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero). | 1 year
  Difference in pain distribution in terms of Hip injury and Osteoarthritis Outcome Score (HOOS) in patients with possible neuropathic pain (neuropathic pain score above 3) and patients without any kind of neuropathic pain (score equal to zero).

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Østerbro, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided